CLINICAL TRIAL: NCT00609167
Title: A Phase II Trial of Cyclophosphamide, Bortezomib and Dexamethasone (CYBOR-D) in Patients With Newly Diagnosed Active Multiple Myeloma
Brief Title: Cyclophosphamide, Bortezomib, and Dexamethasone in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Alexander Keith Stewart, M.B.Ch.B, Mayo Clinic Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000583225; P30CA015083 (NIH); MC0686 (Other: Macyo Clinic Cancer Center); 06-002613 (Other: Mayo Clinic IRB); NCI-2010-02147 (Registry Identifier: NCI-CTRP)
Record Dates: First submitted 2008-01-31; First posted 2008-02-06 (Estimated); Results first posted 2010-12-07 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bortezomib — First 33 patients: 1.3 mg/m^2 IV Days 1, 4, 8 & 11
  Remaining 30 patients: 1.5 mg/m^2 IV Days 1, 8, 15 & 22
Drug: cyclophosphamide — 300mg/m^2 PO days 1, 8, 15 & 22
Drug: dexamethasone — First 33 patients: 40 mg PO Days 1-4, 9-12, 17-20
  Remaining 30 patients: 40 mg PO Days 1-4, 9-12, 17-20 for cycles 1-2; Days 1, 8, 15, 22 for cycle 3+2 for cycle 3 and beyond

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as cyclophosphamide and dexamethasone work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving cyclophosphamide and dexamethasone together with bortezomib may kill more cancer cells.

PURPOSE: This phase II trial is studying giving cyclophosphamide and dexamethasone together with bortezomib to see how well it works in treating patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the response rate (complete response [CR], near CR [nCR], and very good partial response) in patients with newly diagnosed multiple myeloma treated with bortezomib in combination with cyclophosphamide and dexamethasone .

Secondary

* Determine the overall response rate (partial response, PR, or better) in these patients after 4, 8, and 12 courses of this regimen.
* Determine the duration of progression-free and overall survival of patients treated with this regimen.
* To evaluate the toxicity of this regimen in these patients.
* To evaluate the ability to successfully collect peripheral blood stem cells from these patients after 4 months of this regimen.
* To evaluate the CR or nCR rate in these patients after 8 and 12 courses of this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral cyclophosphamide on days 1, 8, 15, and 22; bortezomib IV on days 1, 4, 8 , and 11 OR days 1, 8, 15 and 22; and dexamethasone on days 1-4, 9-12, and 17-20 in courses 1 and 2 and days 1, 18, 15, and 22 in all subsequent courses. Courses repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of symptomatic multiple myeloma

  * Durie Salmon stage 2 or higher
  * Previously untreated multiple myeloma (including immunomodulatory drugs such as thalidomide) with the exception of bisphosphonates
* Evaluable or measurable disease, as defined by at least one of the following:

  * Serum monoclonal protein ≥ 1 g/dL (measurable disease)
  * Urine monoclonal protein ≥ 200 mg/24 hours by protein electrophoresis (measurable disease)
  * Serum-free light chains (FLC) ≥ 10 mg/dL, kappa or lambda, accompanied by an abnormal kappa/lambda ratio

Serum FLC's should only be used for patients without measurable serum or urine m-spike

- Monoclonal bone marrow plasmacytosis ≥ 30% (evaluable disease)

* Patients diagnosed with smoldering myeloma or monoclonal gammopathy of undetermined significance are not eligible

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0, 1, or 2

  - ECOG PS of 3 will be allowed if secondary to pain in the opinion of the Investigator
* Total bilirubin normal OR direct bilirubin ≤ 2.0 mg/dL
* Alkaline phosphatase ≤ 3 times upper limit of normal (ULN)
* AST ≤ 3 times ULN
* Creatinine ≤ 3.5 mg/dL
* Absolute neutrophil count ≥ 1,000/mm³ without transfusion or growth factor
* Platelet count ≥ 100,000/mm³ without transfusion or growth factor
* Willingness and the physical and mental capability to provide written informed consent
* Willingness to return to Mayo Clinic Arizona/Princess Margaret Hospital for follow-up
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion criteria:

* Peripheral sensory neuropathy ≥ grade 2 as defined by National Cancer Institute (NCI) Common Terminology for Common Adverse Events (CTCAE) version 3.0
* Known hypersensitivity to compounds containing boron or mannitol
* Active uncontrolled infection
* Severe cardiac comorbidity including but not limited to:

  * New York Heart Association class III or IV heart failure
  * History of myocardial infarction within the past 6 months
  * Uncontrolled angina or electrocardiographic (ECG) evidence of acute ischemia
  * Severe uncontrolled ventricular arrhythmias or ECG evidence of active conduction system abnormalities
  * Cardiac amyloidosis with hypotension (i.e., systolic blood pressure < 100 mm Hg)
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent study compliance or completion of study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior high-dose corticosteroid therapy for 12 days or less is permitted for emergent complications from newly diagnosed multiple myeloma
* More than 14 days since prior investigational agents
* No concurrent steroids or any other anticancer agents or treatments

  - Patients may receive the equivalent of up to 20 mg prednisone per day for concurrent illness or adrenal replacement therapy
* Concurrent palliative radiotherapy for bony pain or fracture is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-12; Primary Completion 2009-01 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Keith Stewart, M.B., Ch.B., Principal Investigator — Mayo Clinic
Locations (2):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Reeder CB, Reece DE, Kukreti V, Chen C, Trudel S, Hentz J, Noble B, Pirooz NA, Spong JE, Piza JG, Zepeda VH, Mikhael JR, Leis JF, Bergsagel PL, Fonseca R, Stewart AK. Cyclophosphamide, bortezomib and dexamethasone induction for newly diagnosed multiple myeloma: high response rates in a phase II clinical trial. Leukemia. 2009 Jul;23(7):1337-41. doi: 10.1038/leu.2009.26. Epub 2009 Feb 19. PMID 19225538
- [Result] Reeder CB, Reece DE, Kukreti V, Chen C, Trudel S, Laumann K, Hentz J, Pirooz NA, Piza JG, Tiedemann R, Mikhael JR, Bergsagel PL, Leis JF, Fonseca R, Stewart AK. Once- versus twice-weekly bortezomib induction therapy with CyBorD in newly diagnosed multiple myeloma. Blood. 2010 Apr 22;115(16):3416-7. doi: 10.1182/blood-2010-02-271676. No abstract available. PMID 20413666

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-three(63) participants were recruited between December 2006 and October 2008 at either Mayo Clinic Arizona or Princess Margaret Hospital.
Groups:
- CyBorD (Bortezomib 1.3mg/m^2): Bortezomib 1.3mg/m^2 by IV days 1, 4, 8 & 11
  Cyclophosphamide 300mg/m^2 PO days 1, 8, 15 & 22
  Dexamethasone 40mg PO days 1-4, 9-12, 17-20
- CyBorD (Bortezomib 1.5mg/m^2): Bortezomib 1.5mg/m^2 by IV days 1, 8, 15 & 22
  Cyclophosphamide 300mg/m^2 PO days 1, 8, 15 & 22
  Dexamethasone 40mg PO cycle 1-2 days 1-4, 9-12, 17-20, cycle 3 and beyond days 1, 8, 15 & 22
Period: Overall Study
Arm/Group | CyBorD (Bortezomib 1.3mg/m^2) | CyBorD (Bortezomib 1.5mg/m^2)
Started | 33 | 30
Completed | 25 | 23
Not Completed | 8 | 7
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 5 | 1
Not completed — Disease Progression | 1 | 0
Not completed — Stem Cell Transplant | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CyBorD (Bortezomib 1.3mg/m^2) | CyBorD (Bortezomib 1.5mg/m^2) | Total
Number analyzed (Participants) | 33 | 30 | 63
Age Continuous [Median (Full Range); unit: years] | 60 [38 to 75] | 61 [36 to 70] | 61 [36 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 17 | 16 | 33
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
  Canada | 21 | 18 | 39
Parameters of Hematologic Response - Serum M-spike >=1g/dL [Number; unit: participants]
  Yes | 25 | 18 | 43
  No | 8 | 12 | 20
Parameter of Hematologic Response - Serum Immunoglobulin Free Light Chain >=10mg/dL [Number; unit: participants]
  Yes | 24 | 26 | 50
  No | 9 | 4 | 13
Parameter of Hematologic Response - Urine M-Spike >= 200mg/24 hours [Number; unit: participants]
  Yes | 16 | 11 | 27
  No | 17 | 19 | 36
Parameter of Hematologic Response - Bone Marrow Plasma Cells > 30% [Number; unit: participants]
  Yes | 23 | 22 | 45
  No | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a Confirmed Responses Defined as a Complete Response (CR), Near CR or Very Good Partial Response (VGPR) After the First 4 Months of Treatment
Description: Response that was confirmed on 2 consecutive evaluations during the first 4 months of treatment.
  Complete Response(CR): Complete disappearance of M-protein from serum and urine on immunofixation, normalization of Free Light Chain (FLC) ratio and <5% plasma cells in bone marrow.
  near Complete Response (nCR): Patients who meet all criteria for CR except a positive immunofixation will be classified as nCR.
  Very Good Partial Response(VGPR): >=90% reduction in serum M-component; Urine M-Component <100mg per 24hours; <=5% plasma cells in bone marrow.
Time Frame: After 4 months of treatment
Measure: Number; unit: participants
Arm/Group | CyBorD (Bortezomib 1.3mg/m^2) | CyBorD (Bortezomib 1.5mg/m^2)
Number analyzed (Participants) | 33 | 30
participants | 20 | 18

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from registration to progression or death due to any cause.
  Progression was defined as any one or more of the following:
  An increase of 25% from lowest confirmed response in:
  * Serum M-component (absolute increase >= 0.5g/dl)
  * Urine M-component (absolute increase >= 200mg/24hour
  * Difference between involved and uninvolved Free Light Chain levels (absolute increase >= 10mg/dl)
  * Bone marrow plasma cell percentage (absolute increase of >=10%)
  * Definite development of new bone lesion or soft tissue plasmacytomas
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CyBorD (Bortezomib 1.3mg/m^2) | CyBorD (Bortezomib 1.5mg/m^2)
Number analyzed (Participants) | 33 | 30
months | NA [NA to NA] — The median PFS for group 1 has not been attained. | NA [NA to NA] — The median PFS for group 2 has not been attained

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from registration to death of any cause.
Time Frame: From date of registration until death (up to 5 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CyBorD (Bortezomib 1.3mg/m^2) | CyBorD (Bortezomib 1.5mg/m^2)
Number analyzed (Participants) | 33 | 30
months | NA [NA to NA] — Median OS for group 1 has not been attained. | NA [NA to NA] — Median OS for group 2 has not been attained.

4. Secondary Outcome: Number of Participants Who Responded to Treatment (Complete Response,CR; Near Complete Response, nCR; Very Good Partial Response, VGPR; or Partial Response, PR) After 4 Cycles
Description: Response that was confirmed on 2 consecutive evaluations after 8 months of treatment.
  CR, nCR and VGPR as defined in the primary outcome.
  Partial Response(PR): >=50% reduction in serum M-component and/or
  Urine M-Component >=90% reduction or <200mg per 24hours; or >=50% decrease in difference between involved and uninvolved FLC levels.
Time Frame: 4 cycles
Population: Participants who received 4 cycles of treatment were analyzed.
Measure: Number; unit: participants
Arm/Group | CyBorD (Bortezomib 1.3mg/m^2) | CyBorD (Bortezomib 1.5mg/m^2)
Number analyzed (Participants) | 33 | 30
participants | 29 | 28

5. Secondary Outcome: Duration of Response
Description: Duration of response was calculated from the documentation (date) of first response (CR, nCR, VGPR, or PR) until the date of progression or last follow-up in the subset of patients who responded.
Time Frame: Duration of study (up to 12 cycles)
Population: Participants who achieved a partial response(PR) or better were evaluable for this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CyBorD (Bortezomib 1.3mg/m^2) | CyBorD (Bortezomib 1.5mg/m^2)
Number analyzed (Participants) | 29 | 28
months | NA [NA to NA] — Median duration of response for group 1 was not attained. | NA [NA to NA] — Median duration of response for group 2 was not attained.

6. Secondary Outcome: Number of Participants Who Responded to Treatment (CR, nCR, VGPR or PR) After 8 Cycles
Description: Response that was confirmed on 2 consecutive evaluations after 8 cycles of treatment.
  Criteria for CR, nCR, VGPR and PR are defined in prior outcomes.
Time Frame: After 8 cycles of treatment
Population: Participants who received 8 cycles of treatment were analyzed.
Measure: Number; unit: participants
Arm/Group | CyBorD (Bortezomib 1.3mg/m^2) | CyBorD (Bortezomib 1.5mg/m^2)
Number analyzed (Participants) | 0 | 2
participants |  | 1

7. Secondary Outcome: Number of Participants Who Responded to Treatment (CR, nCR, VGPR or PR) After 12 Cycles
Description: Response that was confirmed on 2 consecutive evaluations after 12 cycles of treatment.
  Criteria for CR, nCR, VGPR and PR are defined in prior outcomes.
Time Frame: After 12 cycles of treatment
Population: No participants received 12 cycles of treatment; therefore, all participants are non-evalualble.
Measure: Number; unit: participants
Arm/Group | CyBorD (Bortezomib 1.3mg/m^2) | CyBorD (Bortezomib 1.5mg/m^2)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Severe Adverse Events
Description: Severe adverse events were defined as grade 3 or higher, regardless of attribution to study drugs. Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.
Time Frame: Every cycle during treatment (up to 12 cycles)
Measure: Number; unit: participants
Arm/Group | CyBorD (Bortezomib 1.3mg/m^2) | CyBorD (Bortezomib 1.5mg/m^2)
Number analyzed (Participants) | 33 | 30
participants | 16 | 11

9. Secondary Outcome: Participants Who Successfully Completed Collection of Peripheral Blood Stem Cells for Transplant
Description: Evaluation of the ability to successfully collect peripheral blood stem cells following four months (cycles) of combination therapy.
Time Frame: After 4 cycles of treatment
Population: At the time of publication, data was available on 18 patients for group 2.
Measure: Number; unit: participants
Arm/Group | CyBorD (Bortezomib 1.3mg/m^2) | CyBorD (Bortezomib 1.5mg/m^2)
Number analyzed (Participants) | 33 | 18
participants | 33 | 17

ADVERSE EVENTS:
Arm/Group | CyBorD (Bortezomib 1.3mg/m^2) | CyBorD (Bortezomib 1.5mg/m^2)
Serious Adverse Events (participants affected / at risk) | 4/33 | 3/30
Other Adverse Events (participants affected / at risk) | 33/33 | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CyBorD (Bortezomib 1.3mg/m^2) (N=33) | CyBorD (Bortezomib 1.5mg/m^2) (N=30)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood Infection (Infections and infestations) | 1 (1) | 0 (0)
Lung (pneumonia) infection (Infections and infestations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CyBorD (Bortezomib 1.3mg/m^2) (N=33) | CyBorD (Bortezomib 1.5mg/m^2) (N=30)
Anemia (Blood and lymphatic system disorders) | 4 (6) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 2 (4)
Ischemia/Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 3 (4)
Fatigue (General disorders) | 18 (52) | 24 (75)
Bronchus infection (Infections and infestations) | 0 (0) | 1 (1)
Conjunctiva infection (Infections and infestations) | 0 (0) | 1 (1)
Infection without neutropenia (Infections and infestations) | 0 (0) | 1 (1)
Upper airway infection (Infections and infestations) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Metabolic/Lab (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 14 (30) | 7 (16)
Platelet count decreased (Investigations) | 27 (68) | 11 (28)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (7) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 21 (52) | 17 (64)
Taste (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Euphoria (Psychiatric disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (4) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes